CLINICAL TRIAL: NCT00864474
Title: DRUG USE INVESTIGATION FOR HIV INFECTION PATIENTS OF MARAVIROC (REGULATORY POST MARKETING COMMITMENT PLAN).
Brief Title: Safety And Efficacy Of Maraviroc In Patients For HIV Patients (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4001093
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: CCR5-tropic HIV-1 Infection
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Maraviroc Tablets: Patients administered.
  Interventions: Drug: CELSENTRI® Tablets

INTERVENTIONS:
Drug: CELSENTRI® Tablets — CELSENTRI ® Tablets 150mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dosage is 300 mg twice daily. Maraviroc must be used in combination with other anti-HIV drugs. The dosage may be adjusted according to co-administered medical products. Maraviroc can be taken with or without food".
  Other Names: CELSENTRI® Tablets, maraviroc, Selzentry

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first CELSENTRI® Tablets should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be administered CELSENTRI® Tablets in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not administered CELSENTRI® Tablets.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A4001093 prescribes the Maraviroc Tablets (CELSENTRI® Tablets).
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001093&StudyName=Safety%20And%20Efficacy%20Of%20Maraviroc%20In%20Patients%20For%20HIV%20Patients%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Celsentri (Maraviroc) Tablets: Human immunodeficiency virus (HIV) infected participants, prescribed with Celsentri tablet 150 milligram (mg) depending upon physician's discretion, within the duration from April 2009 to March 2017 were enrolled in the study. Frequency and duration of taking Celsentri tablet were according to package insert, "The usual adult dosage is 300 mg twice daily. Maraviroc must be used in combination with other anti-HIV drugs. The dosage may be adjusted according to co-administered medical products. Maraviroc can be taken with or without food". The participants in this study were retrospectively observed from the first dosing date of Celsentri tablet to the completion of study or treatment discontinuation due to reasons such as participant's death or hospital transfer, within the duration from April 2009 to December 2018.
Period: Overall Study
Arm/Group | Celsentri (Maraviroc) Tablets
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants those who were registered in this study from April 1, 2009 to March 31, 2017.
Groups:
- Celsentri (Maraviroc) Tablets: HIV infected participants, prescribed with Celsentri tablet 150 mg depending upon physician's discretion, within the duration from April 2009 to March 2017 were enrolled in the study. Frequency and duration of taking Celsentri tablet were according to package insert, "The usual adult dosage is 300 mg twice daily. Maraviroc must be used in combination with other anti-HIV drugs. The dosage may be adjusted according to co-administered medical products. Maraviroc can be taken with or without food". The participants in this study were retrospectively observed from the first dosing date of Celsentri tablet to the completion of study or treatment discontinuation due to reasons such as participant's death or hospital transfer, within the duration from April 2009 to December 2018.
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.31 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 67
  Others | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs)
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants | 23.53

2. Primary Outcome: Number of Participants With Unknown Adverse Drug Reactions (ADRs)
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. Unknown ADRs were the ADRs those were not listed on the package insert.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
Participants | 8

3. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Gender
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by gender are reported to assess gender as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, number analyzed ('n') signifies participants who were evaluable for this outcome measure as per gender.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Males: number analyzed (Participants) | 65
  Males | 23.08
  Females: number analyzed (Participants) | 3
  Females | 33.33

4. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Age
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by age are reported to assess age as a risk factor for ADR. ">=" refers to greater than or equal to.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per age.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  >=15 and less than(<) 65 years: number analyzed (Participants) | 63
  >=15 and less than(<) 65 years | 22.22
  >=65 and less than or equal to (<=) 70 years: number analyzed (Participants) | 5
  >=65 and less than or equal to (<=) 70 years | 40.00

5. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Inpatient or Outpatient Status
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by inpatient or outpatient status are reported to assess inpatient or outpatient status as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per inpatient or outpatient status.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Inpatient: number analyzed (Participants) | 2
  Inpatient | 0.00
  Outpatient: number analyzed (Participants) | 45
  Outpatient | 15.56
  Inpatient and outpatient: number analyzed (Participants) | 21
  Inpatient and outpatient | 42.86

6. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Ethnicity
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by ethnicity are reported to assess ethnicity as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per ethnicity.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Japanese: number analyzed (Participants) | 67
  Japanese | 23.88
  Others: number analyzed (Participants) | 1
  Others | 0.00

7. Primary Outcome: Primary: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of History of Therapies for Human Immuno-Deficiency Virus (HIV) Infection
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of history of therapies for HIV Infection are reported to assess presence or absence of history of therapies for HIV Infection as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of history of therapies for HIV Infection.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  History of Therapies for HIV Infection: Absent: number analyzed (Participants) | 16
  History of Therapies for HIV Infection: Absent | 18.75
  History of Therapies for HIV Infection: Present: number analyzed (Participants) | 52
  History of Therapies for HIV Infection: Present | 25.00

8. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor HIV Infection Duration
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by HIV infection duration are reported to assess HIV infection duration as a risk factor for ADR. Unknown: participants for which the duration of HIV infection was not known.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per duration of HIV infection.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  <=1 year: number analyzed (Participants) | 1
  <=1 year | 0.00
  greater than (>) 4 and <=5 years: number analyzed (Participants) | 1
  greater than (>) 4 and <=5 years | 0.00
  >5 years: number analyzed (Participants) | 4
  >5 years | 50.00
  Unknown: number analyzed (Participants) | 62
  Unknown | 22.58

9. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of Allergies
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of allergies are reported to assess presence or absence of allergies as a risk factor for ADR. Unknown: participants for which the presence or absence of allergies was not known.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of allergies.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Allergies: Absent: number analyzed (Participants) | 54
  Allergies: Absent | 18.52
  Allergies: Present: number analyzed (Participants) | 13
  Allergies: Present | 38.46
  Allergies: Unknown: number analyzed (Participants) | 1
  Allergies: Unknown | 100.00

10. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of Comorbidities
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of comorbidities are reported to assess presence or absence of comorbidities as a risk factor for ADR. Comorbidity referred to the presence of co-existing or additional diseases along with HIV infection.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of comorbidities.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Comorbidities: Absent: number analyzed (Participants) | 13
  Comorbidities: Absent | 15.38
  Comorbidities: Present: number analyzed (Participants) | 55
  Comorbidities: Present | 25.45

11. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of Renal Impairment
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of renal impairment are reported to assess presence or absence of renal impairment as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of renal impairment.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Renal Impairment: Absent: number analyzed (Participants) | 62
  Renal Impairment: Absent | 20.97
  Renal Impairment: Present: number analyzed (Participants) | 6
  Renal Impairment: Present | 50.00

12. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of Hepatic Impairment
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of hepatic impairment are reported to assess presence or absence of hepatic impairment as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of hepatic impairment.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Hepatic Impairment: Absent: number analyzed (Participants) | 46
  Hepatic Impairment: Absent | 21.74
  Hepatic Impairment: Present: number analyzed (Participants) | 22
  Hepatic Impairment: Present | 27.27

13. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of Hemophilia
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of hemophilia are reported to assess presence or absence of hemophilia as a risk factor for ADR. Hemophilia is a bleeding disorder that slows the blood clotting process. Participants with this condition experience prolonged bleeding or oozing following an injury, surgery, or having a tooth pulled.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of hemophilia.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Hemophilia: Absent: number analyzed (Participants) | 61
  Hemophilia: Absent | 22.95
  Hemophilia: Present: number analyzed (Participants) | 7
  Hemophilia: Present | 28.57

14. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Mean Daily Dose of Celsentri
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by mean daily dose of Celsentri are reported to assess mean daily dose of Celsentri as a risk factor for ADR. One tablet of Celsentri had a dose of 150 mg.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per mean daily dose of Celsentri.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  <2 tablets: number analyzed (Participants) | 4
  <2 tablets | 0
  2 tablets: number analyzed (Participants) | 36
  2 tablets | 16.67
  >2 tablets: number analyzed (Participants) | 28
  >2 tablets | 35.71

15. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Number of Concomitant Anti-HIV Drugs Use
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by number of concomitant anti-HIV treatment are reported to assess number of concomitant anti-HIV treatment as a risk factor for ADR. Concomitant drugs refers to the drugs other than Celsentri.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per number of concomitant anti-HIV treatments use.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  1 drug: number analyzed (Participants) | 5
  1 drug | 0.00
  2 drugs: number analyzed (Participants) | 17
  2 drugs | 23.53
  3 drugs: number analyzed (Participants) | 28
  3 drugs | 25.00
  >=4 drugs: number analyzed (Participants) | 18
  >=4 drugs | 27.78

16. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Centers for Disease Control and Prevention (CDC) Classification
Description: An ADR:any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by physician.Participants are divided into 3 categories as per CDC classification based on level of HIV infection: Category A= asymptomatic HIV-1 infection, persistent generalized lymphadenopathy and acute(primary)HIV-1 infection with accompanying illness or history of acute HIV-1 infection in adult or adolescent aged>=13 years, Category B: conditions attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or the conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection in an HIV-infected adolescent or adult; and Category C: clinical conditions listed in the acquired immunodeficiency syndrome (AIDS) diagnostic criteria, corresponding to conventional AIDS. Unknown: Participants for which CDC classification was not described.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per CDC classification.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  CDC category A: number analyzed (Participants) | 29
  CDC category A | 20.69
  CDC category B: number analyzed (Participants) | 5
  CDC category B | 20.00
  CDC category C: number analyzed (Participants) | 31
  CDC category C | 29.03
  Unknown: number analyzed (Participants) | 3
  Unknown | 0.00

17. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor as Per Presence or Absence of Concomitant Therapies
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of concomitant therapies are reported to assess presence or absence of concomitant therapies as a risk factor for ADR. Concomitant therapies were the treatments taken by participants to treat comorbid conditions.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of concomitant therapies.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  Concomitant Therapies: Absent: number analyzed (Participants) | 55
  Concomitant Therapies: Absent | 20.00
  Concomitant Therapies: Present: number analyzed (Participants) | 13
  Concomitant Therapies: Present | 38.46

18. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Presence or Absence of Use of Cytochrome P450 3A4 (CYP3A4) Enzyme Inducer Taken Along With Celsentri
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by presence or absence of concomitant CYP3A4 enzyme inducer use are reported to assess presence or absence of concomitant CYP3A enzyme inducer use as a risk factor for ADR. CYP3A4 is an important enzyme in the body, mainly found in the liver and in the intestine. This enzyme is responsible for metabolism of majority of drugs. Many of the food substances and commonly used drugs act as inducer for enzyme CYP3A4.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per presence or absence of concomitant CYP3A enzyme inducer use.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  CYP3A Enzyme Inducer Use: Absent: number analyzed (Participants) | 55
  CYP3A Enzyme Inducer Use: Absent | 21.82
  CYP3A Enzyme Inducer Use: Present: number analyzed (Participants) | 13
  CYP3A Enzyme Inducer Use: Present | 30.77

19. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Total Number of Days of Administration of Celsentri
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by total number of days of administration of Celsentri are reported to assess total number of days of administration of Celsentri as a risk factor for ADR.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per total number of days of administration of Celsentri.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  2 to <=180 days | 8.82
  > 180 and <=365 days: number analyzed (Participants) | 60
  > 180 and <=365 days | 1.67
  > 365 and <=730 days: number analyzed (Participants) | 52
  > 365 and <=730 days | 7.69
  > 730 and <= 2704 days: number analyzed (Participants) | 35
  > 730 and <= 2704 days | 8.57

20. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs): Factor Mean Total Dose of Celsentri
Description: An ADR was any untoward medical occurrence attributed to Celsentri tablets in a participant who received Celsentri tablets. Relatedness to Celsentri tablets was assessed by the physician. In this outcome measure percentage of participants with ADRs categorized by mean total dose of Celsentri are reported to assess mean total dose of Celsentri as a risk factor for ADR. One tablet of Celsentri had a dose of 150 mg.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment. Here, 'n' signifies participants who were evaluable for this outcome measure as per mean total dose of Celsentri.
Measure: Number; unit: percentage of participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
percentage of participants
  4 to <=360 tablets | 7.35
  > 360 and <=730 tablets: number analyzed (Participants) | 61
  > 360 and <=730 tablets | 3.28
  > 730 and <=1460 tablets: number analyzed (Participants) | 53
  > 730 and <=1460 tablets | 0.00
  > 1460 and <=21632 tablets: number analyzed (Participants) | 41
  > 1460 and <=21632 tablets | 17.07

21. Primary Outcome: Number of Adverse Drug Reactions (ADRs) Considered to Have Occurred Due to Effect of Celsentri on Immune Function
Description: as for outcome 1
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: as for outcome 1
Measure: Number; unit: ADRs
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
ADRs | 0

22. Primary Outcome: Number of Adverse Drug Reactions (ADRs) Considered to Have Occurred Due to Effect of Celsentri on Hepatic Function
Description: as for outcome 1
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: as for outcome 1
Measure: Number; unit: ADRs
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
ADRs | 3

23. Primary Outcome: Number of Adverse Drug Reactions (ADRs) Considered to Have Occurred Due to Effect of Celsentri on Cardiovascular Effects
Description: as for outcome 1
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The safety analysis set included all participants who met the criteria for participants and were confirmed to have received at least one dose of Celsentri.
Measure: Number; unit: ADRs
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 68
ADRs | 0

24. Secondary Outcome: Mean Number of Plasma Human Immuno-Deficiency Virus-Ribosomal Ribonucleic Acid (HIV-RNA) Copies: Factor Gender
Description: HIV-RNA copy numbers were measured employing the TaqMan assay with the lower limit of detection of 40 copies per milliliter (copies/mL). The reported data for plasma HIV-RNA copies was calculated after logarithmic conversion.
Time Frame: Month 0 (Baseline), 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81 and 84
Population: Efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here, 'n' signifies participants who were evaluable for this measure for individual gender at respective timepoints.
Measure: Mean (Standard Deviation); unit: Log HIV-RNA copies/milliliter(mL)
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
Log HIV-RNA copies/milliliter(mL)
  Males: Month 0 (Baseline): number analyzed (Participants) | 39
  Males: Month 0 (Baseline) | 3.1 (1.7)
  Males: Month 3: number analyzed (Participants) | 22
  Males: Month 3 | 1.9 (1.0)
  Males: Month 6: number analyzed (Participants) | 17
  Males: Month 6 | 1.6 (0.6)
  Males: Month 9: number analyzed (Participants) | 11
  Males: Month 9 | 1.4 (0.3)
  Males: Month 12: number analyzed (Participants) | 10
  Males: Month 12 | 1.9 (0.8)
  Males: Month 15: number analyzed (Participants) | 12
  Males: Month 15 | 1.7 (0.5)
  Males: Month 18: number analyzed (Participants) | 12
  Males: Month 18 | 1.8 (0.7)
  Males: Month 21: number analyzed (Participants) | 6
  Males: Month 21 | 1.9 (0.6)
  Males: Month 24: number analyzed (Participants) | 7
  Males: Month 24 | 1.5 (0.4)
  Males: Month 27: number analyzed (Participants) | 10
  Males: Month 27 | 1.4 (0.3)
  Males: Month 30: number analyzed (Participants) | 3
  Males: Month 30 | 1.7 (0.4)
  Males: Month 33: number analyzed (Participants) | 11
  Males: Month 33 | 1.3 (0.1)
  Males: Month 36: number analyzed (Participants) | 4
  Males: Month 36 | 1.4 (0.2)
  Males: Month 39: number analyzed (Participants) | 8
  Males: Month 39 | 1.4 (0.3)
  Males: Month 42: number analyzed (Participants) | 6
  Males: Month 42 | 1.5 (0.3)
  Males: Month 45: number analyzed (Participants) | 4
  Males: Month 45 | 1.3 (0.0)
  Males: Month 48: number analyzed (Participants) | 4
  Males: Month 48 | 1.3 (0.0)
  Males: Month 51: number analyzed (Participants) | 4
  Males: Month 51 | 1.3 (0.1)
  Males: Month 54: number analyzed (Participants) | 2
  Males: Month 54 | 219.0 (42.4)
  Males: Month 57: number analyzed (Participants) | 2
  Males: Month 57 | 1294.5 (1096.7)
  Males: Month 60: number analyzed (Participants) | 2
  Males: Month 60 | 1.3 (0.0)
  Males: Month 63: number analyzed (Participants) | 2
  Males: Month 63 | 1.3 (0.0)
  Males: Month 66: number analyzed (Participants) | 0
  Males: Month 69: number analyzed (Participants) | 2
  Males: Month 69 | 1.3 (0.0)
  Males: Month 72: number analyzed (Participants) | 0
  Males: Month 75: number analyzed (Participants) | 1
  Males: Month 75 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Males: Month 78: number analyzed (Participants) | 1
  Males: Month 78 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Males: Month 81: number analyzed (Participants) | 0
  Males: Month 84: number analyzed (Participants) | 1
  Males: Month 84 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 0 (Baseline): number analyzed (Participants) | 1
  Females: Month 0 (Baseline) | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 3: number analyzed (Participants) | 1
  Females: Month 3 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 6: number analyzed (Participants) | 0
  Females: Month 9: number analyzed (Participants) | 0
  Females: Month 12: number analyzed (Participants) | 0
  Females: Month 15: number analyzed (Participants) | 1
  Females: Month 15 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 18: number analyzed (Participants) | 0
  Females: Month 21: number analyzed (Participants) | 0
  Females: Month 24: number analyzed (Participants) | 0
  Females: Month 27: number analyzed (Participants) | 0
  Females: Month 30: number analyzed (Participants) | 0
  Females: Month 33: number analyzed (Participants) | 0
  Females: Month 36: number analyzed (Participants) | 0
  Females: Month 39: number analyzed (Participants) | 0
  Females: Month 42: number analyzed (Participants) | 0
  Females: Month 45: number analyzed (Participants) | 0
  Females: Month 48: number analyzed (Participants) | 0
  Females: Month 51: number analyzed (Participants) | 0
  Females: Month 54: number analyzed (Participants) | 0
  Females: Month 57: number analyzed (Participants) | 0
  Females: Month 60: number analyzed (Participants) | 0
  Females: Month 63: number analyzed (Participants) | 0
  Females: Month 66: number analyzed (Participants) | 0
  Females: Month 69: number analyzed (Participants) | 0
  Females: Month 72: number analyzed (Participants) | 0
  Females: Month 75: number analyzed (Participants) | 0
  Females: Month 78: number analyzed (Participants) | 0
  Females: Month 81: number analyzed (Participants) | 0
  Females: Month 84: number analyzed (Participants) | 0

25. Secondary Outcome: Mean Number of Cluster of Differentiation of More Than 4 (CD4+) Lymphocyte Count: Factor Gender
Description: CD4+ Lymphocyte were counted by CD4 cells per cubic millimeter (cells/mm^3). CD4 cells are the white blood cells and act as laboratory marker providing an indication of immune functioning. A higher number is associated with better immune functioning.
Time Frame: as for outcome 24
Population: Efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom info sirmation about number of CD4 or RNA copies was confirmed. Here, 'n' signifies participants who were evaluable for this measure for individual gender at respective timepoints.
Measure: Mean (Standard Deviation); unit: CD4 cells/mm^3
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
CD4 cells/mm^3
  Males: Month 0 (Baseline): number analyzed (Participants) | 39
  Males: Month 0 (Baseline) | 301.2 (244.5)
  Males: Month 3: number analyzed (Participants) | 22
  Males: Month 3 | 318.2 (221.5)
  Males: Month 6: number analyzed (Participants) | 17
  Males: Month 6 | 319.2 (201.2)
  Males: Month 9: number analyzed (Participants) | 11
  Males: Month 9 | 405.7 (197.6)
  Males: Month 12: number analyzed (Participants) | 10
  Males: Month 12 | 384.0 (228.7)
  Males: Month 15: number analyzed (Participants) | 12
  Males: Month 15 | 440.9 (259.2)
  Males: Month 18: number analyzed (Participants) | 12
  Males: Month 18 | 393.3 (244.8)
  Males: Month 21: number analyzed (Participants) | 6
  Males: Month 21 | 464.7 (302.2)
  Males: Month 24: number analyzed (Participants) | 7
  Males: Month 24 | 427.3 (282.6)
  Males: Month 27: number analyzed (Participants) | 10
  Males: Month 27 | 612.4 (308.7)
  Males: Month 30: number analyzed (Participants) | 3
  Males: Month 30 | 376.0 (161.1)
  Males: Month 33: number analyzed (Participants) | 11
  Males: Month 33 | 447.5 (243.0)
  Males: Month 36: number analyzed (Participants) | 4
  Males: Month 36 | 500.5 (175.3)
  Males: Month 39: number analyzed (Participants) | 8
  Males: Month 39 | 554.4 (252.1)
  Males: Month 42: number analyzed (Participants) | 6
  Males: Month 42 | 794.9 (326.4)
  Males: Month 45: number analyzed (Participants) | 4
  Males: Month 45 | 822.8 (429.8)
  Males: Month 48: number analyzed (Participants) | 4
  Males: Month 48 | 603.0 (368.4)
  Males: Month 51: number analyzed (Participants) | 4
  Males: Month 51 | 637.1 (401.5)
  Males: Month 54: number analyzed (Participants) | 2
  Males: Month 54 | 219.0 (42.4)
  Males: Month 57: number analyzed (Participants) | 2
  Males: Month 57 | 1294.5 (1096.7)
  Males: Month 60: number analyzed (Participants) | 2
  Males: Month 60 | 652.0 (711.3)
  Males: Month 63: number analyzed (Participants) | 2
  Males: Month 63 | 445.0 (377.6)
  Males: Month 66: number analyzed (Participants) | 0
  Males: Month 69: number analyzed (Participants) | 2
  Males: Month 69 | 1006.0 (598.2)
  Males: Month 72: number analyzed (Participants) | 0
  Males: Month 75: number analyzed (Participants) | 1
  Males: Month 75 | 969.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Males: Month 78: number analyzed (Participants) | 1
  Males: Month 78 | 787.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Males: Month 81: number analyzed (Participants) | 0
  Males: Month 84: number analyzed (Participants) | 1
  Males: Month 84 | 934.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 0 (Baseline): number analyzed (Participants) | 1
  Females: Month 0 (Baseline) | 335.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 3: number analyzed (Participants) | 1
  Females: Month 3 | 122.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 6: number analyzed (Participants) | 0
  Females: Month 9: number analyzed (Participants) | 0
  Females: Month 12: number analyzed (Participants) | 0
  Females: Month 15: number analyzed (Participants) | 1
  Females: Month 15 | 197.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Females: Month 18: number analyzed (Participants) | 0
  Females: Month 21: number analyzed (Participants) | 0
  Females: Month 24: number analyzed (Participants) | 0
  Females: Month 27: number analyzed (Participants) | 0
  Females: Month 30: number analyzed (Participants) | 0
  Females: Month 33: number analyzed (Participants) | 0
  Females: Month 36: number analyzed (Participants) | 0
  Females: Month 39: number analyzed (Participants) | 0
  Females: Month 42: number analyzed (Participants) | 0
  Females: Month 45: number analyzed (Participants) | 0
  Females: Month 48: number analyzed (Participants) | 0
  Females: Month 51: number analyzed (Participants) | 0
  Females: Month 54: number analyzed (Participants) | 0
  Females: Month 57: number analyzed (Participants) | 0
  Females: Month 60: number analyzed (Participants) | 0
  Females: Month 63: number analyzed (Participants) | 0
  Females: Month 66: number analyzed (Participants) | 0
  Females: Month 69: number analyzed (Participants) | 0
  Females: Month 72: number analyzed (Participants) | 0
  Females: Month 75: number analyzed (Participants) | 0
  Females: Month 78: number analyzed (Participants) | 0
  Females: Month 81: number analyzed (Participants) | 0
  Females: Month 84: number analyzed (Participants) | 0

26. Secondary Outcome: Mean Number of Plasma Human Immuno-Deficiency Virus-Ribosomal Ribonucleic Acid (HIV-RNA) Copies: Factor The Presence or Absence of Comorbidities
Description: HIV-RNA copy numbers were measured employing the TaqMan assay with the lower limit of detection of 40 copies/mL. The reported data for plasma HIV-RNA copies was calculated after logarithmic conversion.
Time Frame: as for outcome 24
Population: The efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here,'n' signifies participants who were evaluable for this measure for presence or absence of comorbidities at respective timepoints.
Measure: Mean (Standard Deviation); unit: Log HIV-RNA copies/mL
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
Log HIV-RNA copies/mL
  Comorbidities-Present: Month 0 (Baseline): number analyzed (Participants) | 30
  Comorbidities-Present: Month 0 (Baseline) | 2.8 (1.7)
  Comorbidities-Present: Month 3: number analyzed (Participants) | 17
  Comorbidities-Present: Month 3 | 1.9 (1.1)
  Comorbidities-Present: Month 6: number analyzed (Participants) | 12
  Comorbidities-Present: Month 6 | 1.8 (0.7)
  Comorbidities-Present: Month 9: number analyzed (Participants) | 8
  Comorbidities-Present: Month 9 | 1.5 (0.3)
  Comorbidities-Present: Month 12: number analyzed (Participants) | 8
  Comorbidities-Present: Month 12 | 2.1 (0.9)
  Comorbidities-Present: Month 15: number analyzed (Participants) | 10
  Comorbidities-Present: Month 15 | 1.6 (0.6)
  Comorbidities-Present: Month 18: number analyzed (Participants) | 11
  Comorbidities-Present: Month 18 | 1.8 (0.7)
  Comorbidities-Present: Month 21: number analyzed (Participants) | 4
  Comorbidities-Present: Month 21 | 2.1 (0.7)
  Comorbidities-Present: Month 24: number analyzed (Participants) | 7
  Comorbidities-Present: Month 24 | 1.5 (0.4)
  Comorbidities-Present: Month 27: number analyzed (Participants) | 6
  Comorbidities-Present: Month 27 | 1.5 (0.4)
  Comorbidities-Present: Month 30: number analyzed (Participants) | 3
  Comorbidities-Present: Month 30 | 1.7 (0.4)
  Comorbidities-Present: Month 33: number analyzed (Participants) | 7
  Comorbidities-Present: Month 33 | 1.3 (0.2)
  Comorbidities-Present: Month 36: number analyzed (Participants) | 3
  Comorbidities-Present: Month 36 | 1.4 (0.3)
  Comorbidities-Present: Month 39: number analyzed (Participants) | 6
  Comorbidities-Present: Month 39 | 1.5 (0.4)
  Comorbidities-Present: Month 42: number analyzed (Participants) | 4
  Comorbidities-Present: Month 42 | 1.6 (0.4)
  Comorbidities-Present: Month 45: number analyzed (Participants) | 2
  Comorbidities-Present: Month 45 | 1.3 (0.0)
  Comorbidities-Present: Month 48: number analyzed (Participants) | 3
  Comorbidities-Present: Month 48 | 1.3 (0.0)
  Comorbidities-Present: Month 51: number analyzed (Participants) | 3
  Comorbidities-Present: Month 51 | 1.4 (0.1)
  Comorbidities-Present: Month 54: number analyzed (Participants) | 2
  Comorbidities-Present: Month 54 | 1.3 (0.0)
  Comorbidities-Present: Month 57: number analyzed (Participants) | 1
  Comorbidities-Present: Month 57 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 60: number analyzed (Participants) | 2
  Comorbidities-Present: Month 60 | 1.3 (0.0)
  Comorbidities-Present: Month 63: number analyzed (Participants) | 1
  Comorbidities-Present: Month 63 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 66: number analyzed (Participants) | 0
  Comorbidities-Present: Month 69: number analyzed (Participants) | 1
  Comorbidities-Present: Month 69 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 72: number analyzed (Participants) | 0
  Comorbidities-Present: Month 75: number analyzed (Participants) | 1
  Comorbidities-Present: Month 75 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 78: number analyzed (Participants) | 1
  Comorbidities-Present: Month 78 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 81: number analyzed (Participants) | 0
  Comorbidities-Present: Month 84: number analyzed (Participants) | 1
  Comorbidities-Present: Month 84 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 0 (Baseline): number analyzed (Participants) | 10
  Comorbidities-Absent: Month 0 (Baseline) | 3.8 (1.6)
  Comorbidities-Absent: Month 3: number analyzed (Participants) | 6
  Comorbidities-Absent: Month 3 | 1.8 (0.3)
  Comorbidities-Absent: Month 6: number analyzed (Participants) | 5
  Comorbidities-Absent: Month 6 | 1.4 (0.2)
  Comorbidities-Absent: Month 9: number analyzed (Participants) | 3
  Comorbidities-Absent: Month 9 | 1.3 (0.0)
  Comorbidities-Absent: Month 12: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 12 | 1.3 (0.0)
  Comorbidities-Absent: Month 15: number analyzed (Participants) | 3
  Comorbidities-Absent: Month 15 | 1.7 (0.4)
  Comorbidities-Absent: Month 18: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 18 | 2.4 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 21: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 21 | 1.5 (0.3)
  Comorbidities-Absent: Month 24: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 27: number analyzed (Participants) | 4
  Comorbidities-Absent: Month 27 | 1.3 (0.0)
  Comorbidities-Absent: Month 30: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 33: number analyzed (Participants) | 4
  Comorbidities-Absent: Month 33 | 1.3 (0.0)
  Comorbidities-Absent: Month 36: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 36 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 39: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 39 | 1.3 (0.0)
  Comorbidities-Absent: Month 42: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 42 | 1.3 (0.0)
  Comorbidities-Absent: Month 45: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 45 | 1.3 (0.0)
  Comorbidities-Absent: Month 48: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 48 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 51: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 51 | 1.3 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 participant only.
  Comorbidities-Absent: Month 54: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 57: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 57 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 60: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 63: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 63 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 66: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 69: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 69 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 72: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 75: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 78: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 81: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 84: number analyzed (Participants) | 0

27. Secondary Outcome: Mean Number of CD4+ Lymphocyte Counts: Fcator The Presence or Absence of Comorbidities
Description: CD4 cells are the white blood cells and act as laboratory marker providing an indication of immune functioning. A higher number is associated with better immune functioning.
Time Frame: as for outcome 24
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: CD4 cells/mm^3
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
CD4 cells/mm^3
  Comorbidities-Present: Month 0 (Baseline): number analyzed (Participants) | 30
  Comorbidities-Present: Month 0 (Baseline) | 294.2 (249.5)
  Comorbidities-Present: Month 3: number analyzed (Participants) | 17
  Comorbidities-Present: Month 3 | 282.0 (205.0)
  Comorbidities-Present: Month 6: number analyzed (Participants) | 12
  Comorbidities-Present: Month 6 | 284.9 (196.2)
  Comorbidities-Present: Month 9: number analyzed (Participants) | 8
  Comorbidities-Present: Month 9 | 361.5 (199.0)
  Comorbidities-Present: Month 12: number analyzed (Participants) | 8
  Comorbidities-Present: Month 12 | 303.3 (170.9)
  Comorbidities-Present: Month 15: number analyzed (Participants) | 10
  Comorbidities-Present: Month 15 | 422.9 (286.3)
  Comorbidities-Present: Month 18: number analyzed (Participants) | 11
  Comorbidities-Present: Month 18 | 401.6 (254.9)
  Comorbidities-Present: Month 21: number analyzed (Participants) | 4
  Comorbidities-Present: Month 21 | 308.4 (221.7)
  Comorbidities-Present: Month 24: number analyzed (Participants) | 7
  Comorbidities-Present: Month 24 | 427.3 (282.6)
  Comorbidities-Present: Month 27: number analyzed (Participants) | 6
  Comorbidities-Present: Month 27 | 558.7 (399.4)
  Comorbidities-Present: Month 30: number analyzed (Participants) | 3
  Comorbidities-Present: Month 30 | 376.0 (161.1)
  Comorbidities-Present: Month 33: number analyzed (Participants) | 7
  Comorbidities-Present: Month 33 | 357.0 (211.6)
  Comorbidities-Present: Month 36: number analyzed (Participants) | 3
  Comorbidities-Present: Month 36 | 415.7 (54.0)
  Comorbidities-Present: Month 39: number analyzed (Participants) | 6
  Comorbidities-Present: Month 39 | 476.4 (243.2)
  Comorbidities-Present: Month 42: number analyzed (Participants) | 4
  Comorbidities-Present: Month 42 | 813.2 (419.6)
  Comorbidities-Present: Month 45: number analyzed (Participants) | 2
  Comorbidities-Present: Month 45 | 1017.5 (579.1)
  Comorbidities-Present: Month 48: number analyzed (Participants) | 3
  Comorbidities-Present: Month 48 | 603.0 (451.2)
  Comorbidities-Present: Month 51: number analyzed (Participants) | 3
  Comorbidities-Present: Month 51 | 714.1 (454.1)
  Comorbidities-Present: Month 54: number analyzed (Participants) | 2
  Comorbidities-Present: Month 54 | 219.0 (42.4)
  Comorbidities-Present: Month 57: number analyzed (Participants) | 1
  Comorbidities-Present: Month 57 | 2070.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 60: number analyzed (Participants) | 2
  Comorbidities-Present: Month 60 | 652.0 (711.3)
  Comorbidities-Present: Month 63: number analyzed (Participants) | 1
  Comorbidities-Present: Month 63 | 178.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 66: number analyzed (Participants) | 0
  Comorbidities-Present: Month 69: number analyzed (Participants) | 1
  Comorbidities-Present: Month 69 | 1429.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 72: number analyzed (Participants) | 0
  Comorbidities-Present: Month 75: number analyzed (Participants) | 1
  Comorbidities-Present: Month 75 | 969.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 78: number analyzed (Participants) | 1
  Comorbidities-Present: Month 78 | 787.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Present: Month 81: number analyzed (Participants) | 0
  Comorbidities-Present: Month 84: number analyzed (Participants) | 1
  Comorbidities-Present: Month 84 | 934.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 0 (Baseline): number analyzed (Participants) | 10
  Comorbidities-Absent: Month 0 (Baseline) | 325.6 (226.1)
  Comorbidities-Absent: Month 3: number analyzed (Participants) | 6
  Comorbidities-Absent: Month 3 | 388.0 (262.5)
  Comorbidities-Absent: Month 6: number analyzed (Participants) | 5
  Comorbidities-Absent: Month 6 | 401.4 (210.1)
  Comorbidities-Absent: Month 9: number analyzed (Participants) | 3
  Comorbidities-Absent: Month 9 | 523.7 (167.4)
  Comorbidities-Absent: Month 12: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 12 | 707.0 (75.0)
  Comorbidities-Absent: Month 15: number analyzed (Participants) | 3
  Comorbidities-Absent: Month 15 | 419.7 (167.0)
  Comorbidities-Absent: Month 18: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 18 | 301.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 21: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 21 | 777.5 (125.2)
  Comorbidities-Absent: Month 24: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 27: number analyzed (Participants) | 4
  Comorbidities-Absent: Month 27 | 693.0 (75.5)
  Comorbidities-Absent: Month 30: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 33: number analyzed (Participants) | 4
  Comorbidities-Absent: Month 33 | 605.8 (234.0)
  Comorbidities-Absent: Month 36: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 36 | 755.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 39: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 39 | 788.5 (55.9)
  Comorbidities-Absent: Month 42: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 42 | 758.5 (17.7)
  Comorbidities-Absent: Month 45: number analyzed (Participants) | 2
  Comorbidities-Absent: Month 45 | 628.0 (258.8)
  Comorbidities-Absent: Month 48: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 48 | 603.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 51: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 51 | 406.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 54: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 57: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 57 | 519.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 60: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 63: number analyzed (Participants) | 1
  Comorbidities-Absent: Month 63 | 712.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 66: number analyzed (Participants) | 0
  Comorbidities -Absent: Month 69: number analyzed (Participants) | 1
  Comorbidities -Absent: Month 69 | 583.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Comorbidities-Absent: Month 72: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 75: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 78: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 81: number analyzed (Participants) | 0
  Comorbidities-Absent: Month 84: number analyzed (Participants) | 0

28. Secondary Outcome: Mean Number of Plasma HIV-RNA Copies: Factor The Centers for Disease Control and Prevention (CDC) Classification
Description: Participants are divided into 3 categories as per CDC classification based on the level of HIV infection as follows: Category A= asymptomatic HIV-1 infection, persistent generalized lymphadenopathy and acute (primary) HIV-1 infection with accompanying illness or history of acute HIV-1 infection in an adult or adolescent aged >=13 years, Category B: conditions attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or the conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection in an HIV-infected adolescent or adult; and Category C: clinical conditions listed in the acquired immunodeficiency syndrome (AIDS) diagnostic criteria, corresponding to conventional AIDS. Once criteria C has occurred, the person will remain in Category C even if symptoms are alleviated.
Time Frame: as for outcome 24
Population: The efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here,'n' signifies participants who were evaluable for this measure for CDC Classification at respective timepoints.
Measure: Mean (Standard Deviation); unit: Log HIV-RNA copies/mL
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
Log HIV-RNA copies/mL
  CDC category A: Month 0 (Baseline): number analyzed (Participants) | 20
  CDC category A: Month 0 (Baseline) | 3.4 (1.7)
  CDC category A: Month 3: number analyzed (Participants) | 13
  CDC category A: Month 3 | 1.6 (0.3)
  CDC category A: Month 6: number analyzed (Participants) | 9
  CDC category A: Month 6 | 1.5 (0.3)
  CDC category A: Month 9: number analyzed (Participants) | 7
  CDC category A: Month 9 | 1.3 (0.2)
  CDC category A: Month 12: number analyzed (Participants) | 5
  CDC category A: Month 12 | 1.5 (0.4)
  CDC category A: Month 15: number analyzed (Participants) | 6
  CDC category A: Month 15 | 1.5 (0.3)
  CDC category A: Month 18: number analyzed (Participants) | 3
  CDC category A: Month 18 | 1.6 (0.6)
  CDC category A: Month 21: number analyzed (Participants) | 2
  CDC category A: Month 21 | 1.5 (0.3)
  CDC category A: Month 24: number analyzed (Participants) | 2
  CDC category A: Month 24 | 1.3 (0.0)
  CDC category A: Month 27: number analyzed (Participants) | 6
  CDC category A: Month 27 | 1.3 (0.0)
  CDC category A: Month 30: number analyzed (Participants) | 0
  CDC category A: Month 33: number analyzed (Participants) | 6
  CDC category A: Month 33 | 1.3 (0.0)
  CDC category A: Month 36: number analyzed (Participants) | 2
  CDC category A: Month 36 | 1.3 (0.0)
  CDC category A: Month 39: number analyzed (Participants) | 3
  CDC category A: Month 39 | 1.3 (0.0)
  CDC category A: Month 42: number analyzed (Participants) | 3
  CDC category A: Month 42 | 1.3 (0.0)
  CDC category A: Month 45: number analyzed (Participants) | 3
  CDC category A: Month 45 | 1.3 (0.0)
  CDC category A: Month 48: number analyzed (Participants) | 2
  CDC category A: Month 48 | 1.3 (0.0)
  CDC category A: Month 51: number analyzed (Participants) | 2
  CDC category A: Month 51 | 1.3 (0.0)
  CDC category A: Month 54: number analyzed (Participants) | 0
  CDC category A: Month 57: number analyzed (Participants) | 1
  CDC category A: Month 57 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 60: number analyzed (Participants) | 0
  CDC category A: Month 63: number analyzed (Participants) | 1
  CDC category A: Month 63 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 66: number analyzed (Participants) | 0
  CDC category A: Month 69: number analyzed (Participants) | 1
  CDC category A: Month 69 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 72: number analyzed (Participants) | 0
  CDC category A: Month 75: number analyzed (Participants) | 1
  CDC category A: Month 75 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 78: number analyzed (Participants) | 1
  CDC category A: Month 78 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 81: number analyzed (Participants) | 0
  CDC category A: Month 84: number analyzed (Participants) | 1
  CDC category A: Month 84 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 0 (Baseline): number analyzed (Participants) | 3
  CDC category B: Month 0 (Baseline) | 1.6 (0.0)
  CDC category B: Month 3: number analyzed (Participants) | 1
  CDC category B: Month 3 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 6: number analyzed (Participants) | 1
  CDC category B: Month 6 | 1.5 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 9: number analyzed (Participants) | 0
  CDC category B: Month 12: number analyzed (Participants) | 0
  CDC category B: Month 15: number analyzed (Participants) | 2
  CDC category B: Month 15 | 2.1 (1.2)
  CDC category B: Month 18: number analyzed (Participants) | 2
  CDC category B: Month 18 | 1.5 (0.3)
  CDC category B: Month 21: number analyzed (Participants) | 0
  CDC category B: Month 24: number analyzed (Participants) | 1
  CDC category B: Month 24 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 27: number analyzed (Participants) | 1
  CDC category B: Month 27 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 30: number analyzed (Participants) | 1
  CDC category B: Month 30 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 33: number analyzed (Participants) | 1
  CDC category B: Month 33 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 36: number analyzed (Participants) | 0
  CDC category B: Month 39: number analyzed (Participants) | 1
  CDC category B: Month 39 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 42: number analyzed (Participants) | 1
  CDC category B: Month 42 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 45: number analyzed (Participants) | 1
  CDC category B: Month 45 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 48: number analyzed (Participants) | 2
  CDC category B: Month 48 | 1.3 (0.0)
  CDC category B: Month 51: number analyzed (Participants) | 1
  CDC category B: Month 51 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 54: number analyzed (Participants) | 0
  CDC category B: Month 57: number analyzed (Participants) | 0
  CDC category B: Month 60: number analyzed (Participants) | 1
  CDC category B: Month 60 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 63: number analyzed (Participants) | 1
  CDC category B: Month 63 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 66: number analyzed (Participants) | 0
  CDC category B: Month 69: number analyzed (Participants) | 0
  CDC category B: Month 72: number analyzed (Participants) | 0
  CDC category B: Month 75: number analyzed (Participants) | 0
  CDC category B: Month 78: number analyzed (Participants) | 0
  CDC category B: Month 81: number analyzed (Participants) | 0
  CDC category B: Month 84: number analyzed (Participants) | 0
  CDC category C: Month 0 (Baseline): number analyzed (Participants) | 17
  CDC category C: Month 0 (Baseline) | 3.0 (1.8)
  CDC category C: Month 3: number analyzed (Participants) | 9
  CDC category C: Month 3 | 2.3 (1.5)
  CDC category C: Month 6: number analyzed (Participants) | 7
  CDC category C: Month 6 | 1.9 (0.9)
  CDC category C: Month 9: number analyzed (Participants) | 4
  CDC category C: Month 9 | 1.6 (0.4)
  CDC category C: Month 12: number analyzed (Participants) | 5
  CDC category C: Month 12 | 2.3 (1.0)
  CDC category C: Month 15: number analyzed (Participants) | 5
  CDC category C: Month 15 | 1.7 (0.4)
  CDC category C: Month 18: number analyzed (Participants) | 7
  CDC category C: Month 18 | 2.0 (0.8)
  CDC category C: Month 21: number analyzed (Participants) | 4
  CDC category C: Month 21 | 2.1 (0.7)
  CDC category C: Month 24: number analyzed (Participants) | 4
  CDC category C: Month 24 | 1.6 (0.4)
  CDC category C: Month 27: number analyzed (Participants) | 3
  CDC category C: Month 27 | 1.8 (0.4)
  CDC category C: Month 30: number analyzed (Participants) | 2
  CDC category C: Month 30 | 1.9 (0.2)
  CDC category C: Month 33: number analyzed (Participants) | 4
  CDC category C: Month 33 | 1.4 (0.2)
  CDC category C: Month 36: number analyzed (Participants) | 2
  CDC category C: Month 36 | 1.5 (0.3)
  CDC category C: Month 39: number analyzed (Participants) | 4
  CDC category C: Month 39 | 1.6 (0.4)
  CDC category C: Month 42: number analyzed (Participants) | 2
  CDC category C: Month 42 | 1.9 (0.3)
  CDC category C: Month 45: number analyzed (Participants) | 0
  CDC category C: Month 48: number analyzed (Participants) | 0
  CDC category C: Month 51: number analyzed (Participants) | 1
  CDC category C: Month 51 | 1.5 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 54: number analyzed (Participants) | 2
  CDC category C: Month 54 | 1.3 (0.0)
  CDC category C: Month 57: number analyzed (Participants) | 1
  CDC category C: Month 57 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 60: number analyzed (Participants) | 1
  CDC category C: Month 60 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 63: number analyzed (Participants) | 0
  CDC category C: Month 66: number analyzed (Participants) | 0
  CDC category C: Month 69: number analyzed (Participants) | 1
  CDC category C: Month 69 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 72: number analyzed (Participants) | 0
  CDC category C: Month 75: number analyzed (Participants) | 0
  CDC category C: Month 78: number analyzed (Participants) | 0
  CDC category C: Month 81: number analyzed (Participants) | 0
  CDC category C: Month 84: number analyzed (Participants) | 0

29. Secondary Outcome: Mean Number of CD4+ Lymphocyte Counts: Factor The Centers for Disease Control and Prevention (CDC) Classification
Description: CD4 cells are the white blood cells and act as a laboratory marker providing an indication of immune functioning. A higher number is associated with better immune functioning. Participants are divided into 3 categories as per CDC classification based on the level of HIV infection as: Category A= asymptomatic HIV-1 infection, persistent generalized lymphadenopathy and acute(primary)HIV-1 infection with accompanying illness or history of acute HIV-1 infection in an adult or adolescent aged>=13 years, Category B: conditions attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or the conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection in an HIV-infected adolescent or adult; and Category C: clinical conditions listed in the AIDS diagnostic criteria, corresponding to conventional AIDS. Once criteria C has occurred, the person will remain in Category C even if symptoms are alleviated.
Time Frame: as for outcome 24
Population: The efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here, 'n' signifies participants who were evaluable for this measure for CDC Classification at respective timepoints.
Measure: Mean (Standard Deviation); unit: CD4 cells/mm^3
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
CD4 cells/mm^3
  CDC category A: Month 0 (Baseline): number analyzed (Participants) | 20
  CDC category A: Month 0 (Baseline) | 347.0 (222.5)
  CDC category A: Month 3: number analyzed (Participants) | 13
  CDC category A: Month 3 | 416.2 (221.9)
  CDC category A: Month 6: number analyzed (Participants) | 9
  CDC category A: Month 6 | 428.3 (175.6)
  CDC category A: Month 9: number analyzed (Participants) | 7
  CDC category A: Month 9 | 457.4 (147.2)
  CDC category A: Month 12: number analyzed (Participants) | 5
  CDC category A: Month 12 | 524.8 (209.5)
  CDC category A: Month 15: number analyzed (Participants) | 6
  CDC category A: Month 15 | 441.2 (183.8)
  CDC category A: Month 18: number analyzed (Participants) | 3
  CDC category A: Month 18 | 401.3 (221.3)
  CDC category A: Month 21: number analyzed (Participants) | 2
  CDC category A: Month 21 | 777.5 (125.2)
  CDC category A: Month 24: number analyzed (Participants) | 2
  CDC category A: Month 24 | 567.5 (307.6)
  CDC category A: Month 27: number analyzed (Participants) | 6
  CDC category A: Month 27 | 784.8 (232.9)
  CDC category A: Month 30: number analyzed (Participants) | 0
  CDC category Month 33: number analyzed (Participants) | 6
  CDC category Month 33 | 531.7 (214.6)
  CDC category A: Month 36: number analyzed (Participants) | 2
  CDC category A: Month 36 | 616.5 (195.9)
  CDC category A: Month 39: number analyzed (Participants) | 3
  CDC category A: Month 39 | 719.3 (126.1)
  CDC category A: Month 42: number analyzed (Participants) | 3
  CDC category A: Month 42 | 617.0 (245.4)
  CDC category A: Month 45: number analyzed (Participants) | 3
  CDC category A: Month 45 | 621.3 (183.4)
  CDC category A: Month 48: number analyzed (Participants) | 2
  CDC category A: Month 48 | 596.0 (9.9)
  CDC category A: Month 51: number analyzed (Participants) | 2
  CDC category A: Month 51 | 609.0 (287.1)
  CDC category A: Month 54: number analyzed (Participants) | 0
  CDC category A: Month 57: number analyzed (Participants) | 1
  CDC category A: Month 57 | 519.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 60: number analyzed (Participants) | 0
  CDC category A: Month 63: number analyzed (Participants) | 1
  CDC category A: Month 63 | 712.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 66: number analyzed (Participants) | 0
  CDC category A: Month 69: number analyzed (Participants) | 1
  CDC category A: Month 69 | 583.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 72: number analyzed (Participants) | 0
  CDC category A: Month 75: number analyzed (Participants) | 1
  CDC category A: Month 75 | 969.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 78: number analyzed (Participants) | 1
  CDC category A: Month 78 | 787.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category A: Month 81: number analyzed (Participants) | 0
  CDC category A : Month 84: number analyzed (Participants) | 1
  CDC category A : Month 84 | 934.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 0 (Baseline): number analyzed (Participants) | 3
  CDC category B: Month 0 (Baseline) | 264.3 (221.4)
  CDC category B: Month 3: number analyzed (Participants) | 1
  CDC category B: Month 3 | 227.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 6: number analyzed (Participants) | 1
  CDC category B: Month 6 | 122.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 9: number analyzed (Participants) | 0
  CDC category B: Month 12: number analyzed (Participants) | 0
  CDC category B: Month 15: number analyzed (Participants) | 2
  CDC category B: Month 15 | 447.5 (337.3)
  CDC category B: Month 18: number analyzed (Participants) | 2
  CDC category B: Month 18 | 371.0 (319.6)
  CDC category B: Month 21: number analyzed (Participants) | 0
  CDC category B: Month 24: number analyzed (Participants) | 1
  CDC category B: Month 24 | 207.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 27: number analyzed (Participants) | 1
  CDC category B: Month 27 | 180.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 30: number analyzed (Participants) | 1
  CDC category B: Month 30 | 218.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 33: number analyzed (Participants) | 1
  CDC category B: Month 33 | 137.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 36: number analyzed (Participants) | 0
  CDC category B: Month 39: number analyzed (Participants) | 1
  CDC category B: Month 39 | 201.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 42: number analyzed (Participants) | 1
  CDC category B: Month 42 | 1221.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 45: number analyzed (Participants) | 1
  CDC category B: Month 45 | 1427.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 48: number analyzed (Participants) | 2
  CDC category B: Month 48 | 610.0 (637.8)
  CDC category B: Month 51: number analyzed (Participants) | 1
  CDC category B: Month 51 | 219.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 54: number analyzed (Participants) | 0
  CDC category B: Month 57: number analyzed (Participants) | 0
  CDC category B: Month 60: number analyzed (Participants) | 1
  CDC category B: Month 60 | 149.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 63: number analyzed (Participants) | 1
  CDC category B: Month 63 | 178.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category B: Month 66: number analyzed (Participants) | 0
  CDC category B: Month 69: number analyzed (Participants) | 0
  CDC category B: Month 72: number analyzed (Participants) | 0
  CDC category B: Month 75: number analyzed (Participants) | 0
  CDC category B: Month 78: number analyzed (Participants) | 0
  CDC category B: Month 81: number analyzed (Participants) | 0
  CDC category B: Month 84: number analyzed (Participants) | 0
  CDC category C: Month 0 (Baseline): number analyzed (Participants) | 17
  CDC category C: Month 0 (Baseline) | 255.9 (268.5)
  CDC category C: Month 3: number analyzed (Participants) | 9
  CDC category C: Month 3 | 165.0 (129.4)
  CDC category C: Month 6: number analyzed (Participants) | 7
  CDC category C: Month 6 | 207.0 (166.7)
  CDC category C: Month 9: number analyzed (Participants) | 4
  CDC category C: Month 9 | 315.3 (264.1)
  CDC category C: Month 12: number analyzed (Participants) | 5
  CDC category C: Month 12 | 243.2 (155.8)
  CDC category C: Month 15: number analyzed (Participants) | 5
  CDC category C: Month 15 | 389.2 (354.3)
  CDC category C: Month 18: number analyzed (Participants) | 7
  CDC category C: Month 18 | 396.1 (276.3)
  CDC category C: Month 21: number analyzed (Participants) | 4
  CDC category C: Month 21 | 308.4 (221.7)
  CDC category C: Month 24: number analyzed (Participants) | 4
  CDC category C: Month 24 | 412.3 (313.9)
  CDC category C: Month 27: number analyzed (Participants) | 3
  CDC category C: Month 27 | 411.7 (224.0)
  CDC category C: Month 30: number analyzed (Participants) | 2
  CDC category C: Month 30 | 455.0 (120.2)
  CDC category C: Month 33: number analyzed (Participants) | 4
  CDC category C: Month 33 | 398.8 (265.6)
  CDC category C: Month 36: number analyzed (Participants) | 2
  CDC category C: Month 36 | 384.5 (3.5)
  CDC category C: Month 39: number analyzed (Participants) | 4
  CDC category C: Month 39 | 519.1 (259.3)
  CDC category C: Month 42: number analyzed (Participants) | 2
  CDC category C: Month 42 | 848.8 (360.3)
  CDC category C: Month 45: number analyzed (Participants) | 0
  CDC category C: Month 48: number analyzed (Participants) | 0
  CDC category C: Month 51: number analyzed (Participants) | 1
  CDC category C: Month 51 | 1111.2 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 54: number analyzed (Participants) | 2
  CDC category C: Month 54 | 219.0 (42.4)
  CDC category C: Month 57: number analyzed (Participants) | 1
  CDC category C: Month 57 | 2070.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 60: number analyzed (Participants) | 1
  CDC category C: Month 60 | 1155.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 63: number analyzed (Participants) | 0
  CDC category C: Month 66: number analyzed (Participants) | 0
  CDC category C: Month 69: number analyzed (Participants) | 1
  CDC category C: Month 69 | 1429.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  CDC category C: Month 72: number analyzed (Participants) | 0
  CDC category C: Month 75: number analyzed (Participants) | 0
  CDC category C: Month 78: number analyzed (Participants) | 0
  CDC category C: Month 81: number analyzed (Participants) | 0
  CDC category C: Month 84: number analyzed (Participants) | 0

30. Secondary Outcome: Mean Number of Plasma HIV-RNA Copies: Factor The Presence or Absence of History of Therapies for HIV Infection
Description: as for outcome 26
Time Frame: as for outcome 24
Population: The efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here, 'n' signifies participants who were evaluable for this measure for presence or absence therapies at respective timepoints.
Measure: Mean (Standard Deviation); unit: Log HIV-RNA copies/mL
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
Log HIV-RNA copies/mL
  Present: Month 0 (Baseline): number analyzed (Participants) | 28
  Present: Month 0 (Baseline) | 2.4 (1.3)
  Present: Month 3: number analyzed (Participants) | 14
  Present: Month 3 | 1.6 (0.4)
  Present: Month 6: number analyzed (Participants) | 12
  Present: Month 6 | 1.7 (0.7)
  Present: Month 9: number analyzed (Participants) | 7
  Present: Month 9 | 1.4 (0.3)
  Present: Month 12: number analyzed (Participants) | 5
  Present: Month 12 | 1.8 (0.5)
  Present: Month 15: number analyzed (Participants) | 11
  Present: Month 15 | 1.6 (0.5)
  Present: Month 18: number analyzed (Participants) | 12
  Present: Month 18 | 1.8 (0.7)
  Present: Month 21: number analyzed (Participants) | 4
  Present: Month 21 | 2.1 (0.5)
  Present: Month 24: number analyzed (Participants) | 6
  Present: Month 24 | 1.5 (0.4)
  Present: Month 27: number analyzed (Participants) | 9
  Present: Month 27 | 1.4 (0.3)
  Present: Month 30: number analyzed (Participants) | 3
  Present: Month 30 | 1.7 (0.4)
  Present: Month 33: number analyzed (Participants) | 10
  Present: Month 33 | 1.3 (0.2)
  Present: Month 36: number analyzed (Participants) | 3
  Present: Month 36 | 1.4 (0.3)
  Present: Month 39: number analyzed (Participants) | 7
  Present: Month 39 | 1.4 (0.3)
  Present: Month 42: number analyzed (Participants) | 5
  Present: Month 42 | 1.5 (0.4)
  Present: Month 45: number analyzed (Participants) | 4
  Present: Month 45 | 1.3 (0.0)
  Present: Month 48: number analyzed (Participants) | 4
  Present: Month 48 | 1.3 (0.0)
  Present: Month 51: number analyzed (Participants) | 4
  Present: Month 51 | 1.3 (0.1)
  Present: Month 54: number analyzed (Participants) | 2
  Present: Month 54 | 1.3 (0.0)
  Present: Month 57: number analyzed (Participants) | 2
  Present: Month 57 | 1.3 (0.0)
  Present: Month 60: number analyzed (Participants) | 2
  Present: Month 60 | 1.3 (0.0)
  Present: Month 63: number analyzed (Participants) | 2
  Present: Month 63 | 1.3 (0.0)
  Present: Month 66: number analyzed (Participants) | 0
  Present: Month 69: number analyzed (Participants) | 2
  Present: Month 69 | 1.3 (0.0)
  Present: Month 72: number analyzed (Participants) | 0
  Present: Month 75: number analyzed (Participants) | 1
  Present: Month 75 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 78: number analyzed (Participants) | 1
  Present: Month 78 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 81: number analyzed (Participants) | 0
  Present: Month 84: number analyzed (Participants) | 1
  Present: Month 84 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 0 (Baseline): number analyzed (Participants) | 12
  Absent: Month 0 (Baseline) | 4.7 (1.4)
  Absent: Month 3: number analyzed (Participants) | 9
  Absent: Month 3 | 2.2 (1.5)
  Absent: Month 6: number analyzed (Participants) | 5
  Absent: Month 6 | 1.6 (0.5)
  Absent: Month 9: number analyzed (Participants) | 4
  Absent: Month 9 | 1.6 (0.3)
  Absent: Month 12: number analyzed (Participants) | 5
  Absent: Month 12 | 2.0 (1.1)
  Absent: Month 15: number analyzed (Participants) | 2
  Absent: Month 15 | 1.7 (0.6)
  Absent: Month 18: number analyzed (Participants) | 0
  Absent: Month 21: number analyzed (Participants) | 2
  Absent: Month 21 | 1.3 (0.0)
  Absent: Month 24: number analyzed (Participants) | 1
  Absent: Month 24 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 27: number analyzed (Participants) | 1
  Absent: Month 27 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 30: number analyzed (Participants) | 0
  Absent: Month 33: number analyzed (Participants) | 1
  Absent: Month 33 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 36: number analyzed (Participants) | 1
  Absent: Month 36 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 39: number analyzed (Participants) | 1
  Absent: Month 39 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 42: number analyzed (Participants) | 1
  Absent: Month 42 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 45: number analyzed (Participants) | 0
  Absent: Month 48: number analyzed (Participants) | 0
  Absent: Month 51: number analyzed (Participants) | 0
  Absent: Month 54: number analyzed (Participants) | 0
  Absent: Month 57: number analyzed (Participants) | 0
  Absent: Month 60: number analyzed (Participants) | 0
  Absent: Month 63: number analyzed (Participants) | 0
  Absent: Month 66: number analyzed (Participants) | 0
  Absent: Month 69: number analyzed (Participants) | 0
  Absent: Month 72: number analyzed (Participants) | 0
  Absent: Month 75: number analyzed (Participants) | 0
  Absent: Month 78: number analyzed (Participants) | 0
  Absent: Month 81: number analyzed (Participants) | 0
  Absent: Month 84: number analyzed (Participants) | 0

31. Secondary Outcome: Mean Number of CD4+ Lymphocyte Counts: Factor Presence or Absence of History of Therapies for HIV Infection
Description: CD4 cells are the white blood cells and act as a laboratory marker providing an indication of immune functioning. A higher number is associated with better immune functioning.
Time Frame: as for outcome 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: CD4 cells/mm^3
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
CD4 cells/mm^3
  Present: Month 0: number analyzed (Participants) | 28
  Present: Month 0 | 334.8 (266.2)
  Present: Month 3: number analyzed (Participants) | 14
  Present: Month 3 | 263.0 (203.8)
  Present: Month 6: number analyzed (Participants) | 12
  Present: Month 6 | 297.6 (214.5)
  Present: Month 9: number analyzed (Participants) | 7
  Present: Month 9 | 393.7 (216.8)
  Present: Month 12: number analyzed (Participants) | 5
  Present: Month 12 | 373.2 (176.2)
  Present: Month 15: number analyzed (Participants) | 11
  Present: Month 15 | 443.2 (240.1)
  Present: Month 18: number analyzed (Participants) | 12
  Present: Month 18 | 393.3 (244.8)
  Present: Month 21: number analyzed (Participants) | 4
  Present: Month 21 | 520.6 (253.8)
  Present: Month 24: number analyzed (Participants) | 6
  Present: Month 24 | 496.2 (236.5)
  Present: Month 27: number analyzed (Participants) | 9
  Present: Month 27 | 607.1 (327.0)
  Present: Month 30: number analyzed (Participants) | 3
  Present: Month 30 | 376.0 (161.1)
  Present: Month 33: number analyzed (Participants) | 10
  Present: Month 33 | 412.1 (224.3)
  Present: Month 36: number analyzed (Participants) | 3
  Present: Month 36 | 540.0 (191.7)
  Present: Month 39: number analyzed (Participants) | 7
  Present: Month 39 | 599.9 (234.2)
  Present: Month 42: number analyzed (Participants) | 5
  Present: Month 42 | 804.7 (363.9)
  Present: Month 45: number analyzed (Participants) | 4
  Present: Month 45 | 822.8 (429.8)
  Present: Month 48: number analyzed (Participants) | 4
  Present: Month 48 | 603.0 (368.4)
  Present: Month 51: number analyzed (Participants) | 4
  Present: Month 51 | 637.1 (401.5)
  Present: Month 54: number analyzed (Participants) | 2
  Present: Month 54 | 219.0 (42.4)
  Present: Month 57: number analyzed (Participants) | 2
  Present: Month 57 | 1294.5 (1096.7)
  Present: Month 60: number analyzed (Participants) | 2
  Present: Month 60 | 652.0 (711.3)
  Present: Month 63: number analyzed (Participants) | 2
  Present: Month 63 | 445.0 (377.6)
  Present: Month 66: number analyzed (Participants) | 0
  Present: Month 69: number analyzed (Participants) | 2
  Present: Month 69 | 1006.0 (598.2)
  Present: Month 72: number analyzed (Participants) | 0
  Present: Month 75: number analyzed (Participants) | 1
  Present: Month 75 | 969.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 78: number analyzed (Participants) | 1
  Present: Month 78 | 787.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 81: number analyzed (Participants) | 0
  Present: Month 84: number analyzed (Participants) | 1
  Present: Month 84 | 934.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 0: number analyzed (Participants) | 12
  Absent: Month 0 | 225.6 (153.5)
  Absent: Month 3: number analyzed (Participants) | 9
  Absent: Month 3 | 382.2 (237.0)
  Absent: Month 6: number analyzed (Participants) | 5
  Absent: Month 6 | 371.0 (175.1)
  Absent: Month 9: number analyzed (Participants) | 4
  Absent: Month 9 | 426.8 (187.7)
  Absent: Month 12: number analyzed (Participants) | 5
  Absent: Month 12 | 394.8 (293.9)
  Absent: Month 15: number analyzed (Participants) | 2
  Absent: Month 15 | 306.5 (430.6)
  Absent: Month 18: number analyzed (Participants) | 0
  Absent: Month 21: number analyzed (Participants) | 2
  Absent: Month 21 | 353.0 (475.2)
  Absent: Month 24: number analyzed (Participants) | 1
  Absent: Month 24 | 14.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 27: number analyzed (Participants) | 1
  Absent: Month 27 | 660.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 30: number analyzed (Participants) | 0
  Absent: Month 33: number analyzed (Participants) | 1
  Absent: Month 33 | 801.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 36: number analyzed (Participants) | 1
  Absent: Month 36 | 382.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 39: number analyzed (Participants) | 1
  Absent: Month 39 | 236.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 42: number analyzed (Participants) | 1
  Absent: Month 42 | 746.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 45: number analyzed (Participants) | 0
  Absent: Month 48: number analyzed (Participants) | 0
  Absent: Month 51: number analyzed (Participants) | 0
  Absent: Month 54: number analyzed (Participants) | 0
  Absent: Month 57: number analyzed (Participants) | 0
  Absent: Month 60: number analyzed (Participants) | 0
  Absent: Month 63: number analyzed (Participants) | 0
  Absent: Month 66: number analyzed (Participants) | 0
  Absent: Month 69: number analyzed (Participants) | 0
  Absent: Month 72: number analyzed (Participants) | 0
  Absent: Month 75: number analyzed (Participants) | 0
  Absent: Month 78: number analyzed (Participants) | 0
  Absent: Month 81: number analyzed (Participants) | 0
  Absent: Month 84: number analyzed (Participants) | 0

32. Secondary Outcome: Mean Number of Plasma HIV-RNA Copies: Factor The Presence or Absence of Use of Cytochrome P450 3A4 (CYP3A4) Enzyme Inducer Taken Along With Celsentri
Description: HIV-RNA copy numbers were measured employing the TaqMan assay with the lower limit of detection of 40 copies/mL. CYP3A4 is an important enzyme in the body, mainly found in the liver and in the intestine. This enzyme is responsible for metabolism of majority of drugs. Many of the food substances and commonly used drugs act as inducers of enzyme CYP3A4. The reported data for plasma HIV-RNA copies was calculated after logarithmic conversion.
Time Frame: as for outcome 24
Population: The efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here, 'n' signifies participants who were evaluable for this measure for presence or absence of CYP3A4 at respective timepoints.
Measure: Mean (Standard Deviation); unit: Log HIV-RNA copies/mL
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
Log HIV-RNA copies/mL
  Present: Month 0 (Baseline): number analyzed (Participants) | 6
  Present: Month 0 (Baseline) | 3.6 (2.4)
  Present: Month 3: number analyzed (Participants) | 5
  Present: Month 3 | 2.4 (2.1)
  Present: Month 6: number analyzed (Participants) | 3
  Present: Month 6 | 1.5 (0.3)
  Present: Month 9: number analyzed (Participants) | 3
  Present: Month 9 | 1.3 (0.0)
  Present: Month 12: number analyzed (Participants) | 1
  Present: Month 12 | 3.9 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 15: number analyzed (Participants) | 4
  Present: Month 15 | 1.6 (0.4)
  Present: Month 18: number analyzed (Participants) | 1
  Present: Month 18 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 21: number analyzed (Participants) | 1
  Present: Month 21 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 24: number analyzed (Participants) | 2
  Present: Month 24 | 1.3 (0.0)
  Present: Month 27: number analyzed (Participants) | 0
  Present: Month 30: number analyzed (Participants) | 0
  Present: Month 33: number analyzed (Participants) | 3
  Present: Month 33 | 1.3 (0.0)
  Present: Month 36: number analyzed (Participants) | 1
  Present: Month 36 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 39: number analyzed (Participants) | 1
  Present: Month 39 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 42: number analyzed (Participants) | 1
  Present: Month 42 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 45: number analyzed (Participants) | 2
  Present: Month 45 | 1.3 (0.0)
  Present: Month 48: number analyzed (Participants) | 1
  Present: Month 48 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 51: number analyzed (Participants) | 2
  Present: Month 51 | 1.3 (0.0)
  Present: Month 54: number analyzed (Participants) | 0
  Present: Month 57: number analyzed (Participants) | 1
  Present: Month 57 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 60: number analyzed (Participants) | 0
  Present: Month 63: number analyzed (Participants) | 1
  Present: Month 63 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 66: number analyzed (Participants) | 0
  Present: Month 69: number analyzed (Participants) | 1
  Present: Month 69 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 72: number analyzed (Participants) | 0
  Present: Month 75: number analyzed (Participants) | 1
  Present: Month 75 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 78: number analyzed (Participants) | 1
  Present: Month 78 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 81: number analyzed (Participants) | 0
  Present: Month 84: number analyzed (Participants) | 1
  Present: Month 84 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 0 (Baseline): number analyzed (Participants) | 34
  Absent: Month 0 (Baseline) | 3.0 (1.6)
  Absent: Month 3: number analyzed (Participants) | 18
  Absent: Month 3 | 1.7 (0.4)
  Absent: Month 6: number analyzed (Participants) | 14
  Absent: Month 6 | 1.7 (0.7)
  Absent: Month 9: number analyzed (Participants) | 8
  Absent: Month 9 | 1.5 (0.3)
  Absent: Month 12: number analyzed (Participants) | 9
  Absent: Month 12 | 1.7 (0.5)
  Absent: Month 15: number analyzed (Participants) | 9
  Absent: Month 15 | 1.6 (0.6)
  Absent: Month 18: number analyzed (Participants) | 11
  Absent: Month 18 | 1.9 (0.7)
  Absent: Month 21: number analyzed (Participants) | 5
  Absent: Month 21 | 2.0 (0.6)
  Absent: Month 24: number analyzed (Participants) | 5
  Absent: Month 24 | 1.6 (0.4)
  Absent: Month 27: number analyzed (Participants) | 10
  Absent: Month 27 | 1.4 (0.3)
  Absent: Month 30: number analyzed (Participants) | 3
  Absent: Month 30 | 1.7 (0.4)
  Absent: Month 33: number analyzed (Participants) | 8
  Absent: Month 33 | 1.3 (0.2)
  Absent: Month 36: number analyzed (Participants) | 3
  Absent: Month 36 | 1.4 (0.3)
  Absent: Month 39: number analyzed (Participants) | 7
  Absent: Month 39 | 1.4 (0.3)
  Absent: Month 42: number analyzed (Participants) | 5
  Absent: Month 42 | 1.5 (0.4)
  Absent: Month 45: number analyzed (Participants) | 2
  Absent: Month 45 | 1.3 (0.0)
  Absent: Month 48: number analyzed (Participants) | 3
  Absent: Month 48 | 1.3 (0.0)
  Absent: Month 51: number analyzed (Participants) | 2
  Absent: Month 51 | 1.4 (0.2)
  Absent: Month 54: number analyzed (Participants) | 2
  Absent: Month 54 | 1.3 (0.0)
  Absent: Month 57: number analyzed (Participants) | 1
  Absent: Month 57 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 60: number analyzed (Participants) | 2
  Absent: Month 60 | 1.3 (0.0)
  Absent: Month 63: number analyzed (Participants) | 1
  Absent: Month 63 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 66: number analyzed (Participants) | 0
  Absent: Month 69: number analyzed (Participants) | 1
  Absent: Month 69 | 1.3 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 72: number analyzed (Participants) | 0
  Absent: Month 75: number analyzed (Participants) | 0
  Absent: Month 78: number analyzed (Participants) | 0
  Absent: Month 81: number analyzed (Participants) | 0
  Absent: Month 84: number analyzed (Participants) | 0

33. Secondary Outcome: Mean Number of CD4+ Lymphocyte: Factor The Presence or Absence of Use of Cytochrome P450 3A4 (CYP3A4) Enzyme Inducer Taken Along With Celsentri
Description: CD4 cells are the white blood cells and act as laboratory marker providing an indication of immune functioning. A higher number is associated with better immune functioning. CYP3A4 is an important enzyme in the body, mainly found in the liver and in the intestine. This enzyme is responsible for metabolism of many of drugs. Many of the food substances and commonly used drugs act as inducers of enzyme CYP3A4.
Time Frame: as for outcome 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: CD4 cells/mm^3
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 63
CD4 cells/mm^3
  Present: Month 0 (Baseline): number analyzed (Participants) | 6
  Present: Month 0 (Baseline) | 200.7 (220.4)
  Present: Month 3: number analyzed (Participants) | 5
  Present: Month 3 | 193.0 (217.3)
  Present: Month 6: number analyzed (Participants) | 3
  Present: Month 6 | 212.0 (233.8)
  Present: Month 9: number analyzed (Participants) | 3
  Present: Month 9 | 223.0 (183.0)
  Present: Month 12: number analyzed (Participants) | 1
  Present: Month 12 | 4.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 15: number analyzed (Participants) | 4
  Present: Month 15 | 231.3 (247.2)
  Present: Month 18: number analyzed (Participants) | 1
  Present: Month 18 | 248.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 21: number analyzed (Participants) | 1
  Present: Month 21 | 17.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 24: number analyzed (Participants) | 2
  Present: Month 24 | 182.0 (237.6)
  Present: Month 27: number analyzed (Participants) | 0
  Present: Month 30: number analyzed (Participants) | 0
  Present: Month 33: number analyzed (Participants) | 3
  Present: Month 33 | 367.7 (29.0)
  Present: Month 36: number analyzed (Participants) | 1
  Present: Month 36 | 478.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 39: number analyzed (Participants) | 1
  Present: Month 39 | 581.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 42: number analyzed (Participants) | 1
  Present: Month 42 | 334.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 45: number analyzed (Participants) | 2
  Present: Month 45 | 526.5 (115.3)
  Present: Month 48: number analyzed (Participants) | 1
  Present: Month 48 | 589.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 51: number analyzed (Participants) | 2
  Present: Month 51 | 609.0 (287.1)
  Present: Month 54: number analyzed (Participants) | 0
  Present: Month 57: number analyzed (Participants) | 1
  Present: Month 57 | 519.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 60: number analyzed (Participants) | 0
  Present: Month 63: number analyzed (Participants) | 1
  Present: Month 63 | 712.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 66: number analyzed (Participants) | 0
  Present: Month 69: number analyzed (Participants) | 1
  Present: Month 69 | 583.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 72: number analyzed (Participants) | 0
  Present: Month 75: number analyzed (Participants) | 1
  Present: Month 75 | 969.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 78: number analyzed (Participants) | 1
  Present: Month 78 | 787.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Present: Month 81: number analyzed (Participants) | 0
  Present: Month 84: number analyzed (Participants) | 1
  Present: Month 84 | 934.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 0 (Baseline): number analyzed (Participants) | 34
  Absent: Month 0 (Baseline) | 320.0 (243.6)
  Absent: Month 3: number analyzed (Participants) | 18
  Absent: Month 3 | 342.1 (215.8)
  Absent: Month 6: number analyzed (Participants) | 14
  Absent: Month 6 | 342.1 (195.4)
  Absent: Month 9: number analyzed (Participants) | 8
  Absent: Month 9 | 474.3 (163.0)
  Absent: Month 12: number analyzed (Participants) | 9
  Absent: Month 12 | 426.2 (197.0)
  Absent: Month 15: number analyzed (Participants) | 9
  Absent: Month 15 | 507.0 (223.5)
  Absent: Month 18: number analyzed (Participants) | 11
  Absent: Month 18 | 406.5 (252.2)
  Absent: Month 21: number analyzed (Participants) | 5
  Absent: Month 21 | 554.3 (232.4)
  Absent: Month 24: number analyzed (Participants) | 5
  Absent: Month 24 | 525.4 (252.0)
  Absent: Month 27: number analyzed (Participants) | 10
  Absent: Month 27 | 612.4 (308.7)
  Absent: Month 30: number analyzed (Participants) | 3
  Absent: Month 30 | 376.0 (161.1)
  Absent: Month 33: number analyzed (Participants) | 8
  Absent: Month 33 | 477.4 (283.5)
  Absent: Month 36: number analyzed (Participants) | 3
  Absent: Month 36 | 508.0 (213.9)
  Absent: Month 39: number analyzed (Participants) | 7
  Absent: Month 39 | 550.6 (272.1)
  Absent: Month 42: number analyzed (Participants) | 5
  Absent: Month 42 | 887.1 (263.5)
  Absent: Month 45: number analyzed (Participants) | 2
  Absent: Month 45 | 1119.0 (435.6)
  Absent: Month 48: number analyzed (Participants) | 3
  Absent: Month 48 | 607.7 (451.0)
  Absent: Month 51: number analyzed (Participants) | 2
  Absent: Month 51 | 665.1 (630.9)
  Absent: Month 54: number analyzed (Participants) | 2
  Absent: Month 54 | 219.0 (42.4)
  Absent: Month 57: number analyzed (Participants) | 1
  Absent: Month 57 | 2070.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 60: number analyzed (Participants) | 2
  Absent: Month 60 | 652.0 (711.3)
  Absent: Month 63: number analyzed (Participants) | 1
  Absent: Month 63 | 178.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 66: number analyzed (Participants) | 0
  Absent: Month 69: number analyzed (Participants) | 1
  Absent: Month 69 | 1429.0 (NA) — Standard deviation could not be calculated since only one participant was available for analysis.
  Absent: Month 72: number analyzed (Participants) | 0
  Absent: Month 75: number analyzed (Participants) | 0
  Absent: Month 78: number analyzed (Participants) | 0
  Absent: Month 81: number analyzed (Participants) | 0
  Absent: Month 84: number analyzed (Participants) | 0

34. Secondary Outcome: Number of Participants With Tropism Switch From CCR5- to CXCR4-Tropic Variants
Description: CCR5= C-C chemokine receptor type 5 and CXCR4= C-X-C chemokine receptor type 4. Tropism switch is the mutation of CCR5-tropic HIV-1 to a CXCR4-using virus.
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Population: The efficacy analysis set included participants infected with HIV, had received Celsentri tablets at least once for HIV as primary indication and in whom information about number of CD4 or RNA copies was confirmed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 32
Participants | 0

35. Secondary Outcome: Mean Number of Plasma HIV-RNA Copies for Participants Who Took Concomitant Therapies Along With Celsentri
Time Frame: as for outcome 24
Population: The efficacy analysis set. Here, "Overall Number of Participants Analyzed" included participants evaluable for this measure. 'n' signifies participants who were evaluable for this measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Log HIV-RNA copies/mL
Arm/Group | Celsentri (Maraviroc) Tablets
Number analyzed (Participants) | 40
Log HIV-RNA copies/mL
  At baseline | 3.1 (1.7)
  At Month 3: number analyzed (Participants) | 23
  At Month 3 | 1.8 (1.0)
  At Month 6: number analyzed (Participants) | 17
  At Month 6 | 1.6 (0.6)
  At Month 9: number analyzed (Participants) | 11
  At Month 9 | 1.4 (0.3)
  At Month 12: number analyzed (Participants) | 10
  At Month 12 | 1.9 (0.8)
  At Month 15: number analyzed (Participants) | 13
  At Month 15 | 1.6 (0.5)
  At Month 18: number analyzed (Participants) | 12
  At Month 18 | 1.8 (0.7)
  At Month 21: number analyzed (Participants) | 6
  At Month 21 | 1.9 (0.6)
  At Month 24: number analyzed (Participants) | 7
  At Month 24 | 1.5 (0.4)
  At Month 27: number analyzed (Participants) | 10
  At Month 27 | 1.4 (0.3)
  At Month 30: number analyzed (Participants) | 3
  At Month 30 | 1.7 (0.4)
  At Month 33: number analyzed (Participants) | 11
  At Month 33 | 1.3 (0.1)
  At Month 36: number analyzed (Participants) | 4
  At Month 36 | 1.4 (0.2)
  At Month 39: number analyzed (Participants) | 8
  At Month 39 | 1.4 (0.3)
  At Month 42: number analyzed (Participants) | 6
  At Month 42 | 1.5 (0.3)
  At Month 45: number analyzed (Participants) | 4
  At Month 45 | 1.3 (0.0)
  At Month 48: number analyzed (Participants) | 4
  At Month 48 | 1.3 (0.0)
  At Month 51: number analyzed (Participants) | 4
  At Month 51 | 1.3 (0.1)
  At Month 54: number analyzed (Participants) | 2
  At Month 54 | 1.3 (0.0)
  At Month 57: number analyzed (Participants) | 2
  At Month 57 | 1.3 (0.0)
  At Month 60: number analyzed (Participants) | 2
  At Month 60 | 1.3 (0.0)
  At Month 63: number analyzed (Participants) | 2
  At Month 63 | 1.3 (0.0)
  At Month 66: number analyzed (Participants) | 0
  At Month 69: number analyzed (Participants) | 2
  At Month 69 | 1.3 (0.0)
  At Month 72: number analyzed (Participants) | 0
  At Month 75: number analyzed (Participants) | 1
  At Month 75 | 1.3 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  At Month 78: number analyzed (Participants) | 1
  At Month 78 | 1.3 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  At Month 81: number analyzed (Participants) | 0
  At Month 84: number analyzed (Participants) | 1
  At Month 84 | 1.3 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

ADVERSE EVENTS:
Time Frame: From April 2009 to December 2018 (up to approximately 8 years 8 months)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another, or a participant may have experienced both a serious and non-serious event. The safety analysis set included participants who were infected with HIV, had received Celsentri tablet at least once and visited physician after first dose of treatment.
Arm/Group | Celsentri (Maraviroc) Tablets
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 17/68
Other Adverse Events (participants affected / at risk) | 20/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celsentri (Maraviroc) Tablets (N=68)
Glaucoma (Eye disorders) | 1
Necrotising retinitis (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1
Aspergillus infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Syphilis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Psychiatric symptom (Psychiatric disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Prerenal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Renal tubular disorder (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celsentri (Maraviroc) Tablets (N=68)
Anaemia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Dermatophytosis of nail (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
White blood cell count increased (Investigations) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT00864474/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT00864474/SAP_001.pdf